CLINICAL TRIAL: NCT05126589
Title: Metagenomic Study on the Distributive Pattern of Respiratory Virus in the Community After the Emergence of COVID-19
Brief Title: Respiratory Virus Metagenomics After COVID-19
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Research Professor, Chinese University of Hong Kong
Other Study IDs: Protocol HK COVID metagenomic
Record Dates: First submitted 2021-11-17; First posted 2021-11-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Respiratory Infection
Keywords: metagenomic; respiratory virus infections; exposure risk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal and throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims to characterize the distributive pattern of viruses in upper airway and its relationship with influenza seasons, symptomatology and exposure setting. A total of 500 adults residing in Hong Kong would be recruited, who would complete a questionnaire and return self-collected nasal and throat swabs for metagenomic analyses.

DETAILED DESCRIPTION:
1. This is a serial cross-sectional study. Participants would be asked to complete a questionnaire and to self-collect nasal and throat swabs during a specified collection period with reference to an influenza season.
2. Subjects would be invited by post through randomly selected households throughout the territory of Hong Kong. Eligible persons are adults normally resident in the address who could communicate in written Chinese or English. Persons incapable of giving informed consent would be excluded. Other exclusion criteria are: individuals with mental illnesses, prisoners. Approval is obtained from the clinical research ethics committee.
3. A bilingual questionnaire would be administered, which consists of four parts, including: (a) Socio-demographics; (b) History of SARS-CoV-1 infection and vaccination; (c) Exposure settings preceding sample collection; (d) Presence and types (if any) of influenza-like illnesses (ILI) at the time of sample collection;
4. With the provision of nasal and throat swab collection kits, participants shall collect the nasal/throat sample within a 3-month period from the start of an influenza season when one presents with influenza-like illnesses (ILI), or at the end of the season if no such illnesses occur. The self-collected swabs would need to be returned with the questionnaire within 48 hours after sampling. After returning the swabs, a HK$50 voucher would be given to compensate participants' time.
5. RNA would be extracted from the collected samples, followed by by metagenomic analyses. The collected data would be tidied, checked and collated to form a research database. Descriptive statistics, including standard frequency tables and metrics, would be performed.
6. The key outcomes in this study are the change of abundance of viruses in different influenza seasons, and the difference in distributions of viral taxa in samples from participants.
7. On completion of the analyses, the transmission risk of respiratory infections could be assessed, and emerging viral infections could be identified. Certain exposure setting associated viruses could be identified to inform public health policies.

ELIGIBILITY:
Inclusion Criteria:

* adults normally residing in Hong Kong
* could communicate in English and/or Chinese
* provision of consent

Exclusion Criteria:

* individuals with mental illness
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects would be invited by post through randomly selected households throughout the territory of Hong Kong.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Positive identification of viruses | 4 years
  Proportion of specimens with identified respiratory virus taxa

CONTACTS AND LOCATIONS:
Overall Officials: Shui Shan Lee, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China